CLINICAL TRIAL: NCT04169672
Title: A Phase II, Open-label, Single-arm, Multi-center Study of the Efficacy and Safety of Surufatinib Single Agent or Surufatinib Combined With Toripalimab in Patients With Advanced Solid Tumors
Brief Title: Study of Surufatinib Single Agent or Surufatinib Combined With Toripalimab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-012-00CH1
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — surufatinib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surufatinib & Toripalimab (Experimental): Surufatinib 250mg will be taken orally once daily continuously through a 21-day cycle of study treatment. Toripalimab 240mg will be intravenously administered on Day 1 of each cycle.
  Interventions: Drug: Surufatinib; Drug: Toripalimab
- Surufatinib (Experimental): Surufatinib 300mg will be taken orally once daily continuously through a 21-day cycle of study treatment.
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Surufatinib is a tablet in the form of 50mg, oral, once a day.
  Other Names: HMPL-012
Drug: Toripalimab — Toripalimab is an injection in the form of 240mg, intravenous, once three weeks.
  Other Names: JS001
  Arms: Surufatinib & Toripalimab

SUMMARY:
This is a phase II, single arm, open-label, multicenter study to evaluate the efficacy and safety of Surufatinib single agent or Surufatinib combined with Toripalimab in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study population is about 260 patients with advanced solid tumors, who fails or can not tolerate standard therapies, or for whom no effective standard therapy is available, or who refuses standard therapies. This study includes two arms. One is that Surufatinib single agent 300mg once a day (QD) will be orally administrated in patients with advanced neuroendocrine carcinoma (NEC). In another arm Surufatinib 250 mg QD will be orally administrated and Toripalimab 240mg will be intravenously administered every 3 weeks up to documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent. For Toripalimab, the upper time limit for treatment is 2 years. The primary objective is safety of safety run-in (about 6 patients) and objective response rate (ORR) of Surufatinib single agent in patients with advanced NEC or Surufatinib combined with Toripalimab in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adequately understand the study and voluntarily sign the Informed Consent Form;
* 18-75 years old;
* Histologically or cytologically confirmed advanced solid tumors (focusing on neuroendocrine neoplasmas (NENs), biliary tract cancer, gastric cancer, thyroid cancer, small cell lung cancer, non-small cell lung cancer, soft tissue sarcoma, endometrial cancer and esophageal squamous cell carcinoma, etc);
* Fail or cannot tolerate the standard therapies, or for whom no effective standard therapy is available, or refuse standard therapy;
* NSCLC cohort: no prior chemotherapy or any other systemic therapy for stage IV NSCLC with positove PD-L1 expression;
* Have a performance status (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale;
* Have measurable lesions (according to RECIST 1.1);
* Agree to provide histology samples;
* Lab tests within 7 days before first dose:

  1. Absolute neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥100×10^9/L, and hemoglobin ≥9 g/dL;
  2. Serum total bilirubin <1.5 times the upper limit of normal (ULN);
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels ≤ 1.5 times the ULN without liver metastases; and ALT and AST ≤ 3 times ULN with liver metastases;
  4. Serum creatinine <1.5 times ULN and creatinine clearance ≥50 mL/min;
  5. Urine protein < 2+; if ≥2+, 24-hour urine protein <1 g;
  6. International Normalized Ratio (INR) ≤1.5 ULN and activated partial thromboplastin time (APTT) ≤1.5 ULN;
* Have expected survival of more than 12 weeks;
* Male or females patients with reproductive potential must agree to use an effective contraceptive method, for example, double-barrier device, condom, oral or injected birth control medication or intrauterine device, during the study and within 90 days after study treatment discontinuation. All female patients are considered to be fertile, unless the patient had natural menopause or artificial menopause or sterilization (such as hysterectomy, bilateral oophorectomy or ovarian irradiation).

Exclusion Criteria:

* Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for hair loss or Grade ≤ 2 peripheral neurotoxicity caused by oxaliplatin);
* Other malignancies diagnosed within the previous 5 years, except skin basal cell carcinoma or skin squamous cell carcinoma or cervical carcinoma in situ;
* Symptomatic central nervous system (CNS) metastasis or cancerous meningitis (meningeal metastasis) during the screening period;
* Systematic anti-tumor therapy received within 4 weeks prior to first dose, including chemotherapy, biotherapy, targeted therapy, hormonotherapy, and anti-tumor Chinese medicine treatment;
* Radical radiotherapy within 4 weeks prior to first dose, radioactive seed implantation within 60 days prior to first dose, or Palliative radiotherapy for a bone metastasis lesion within 1 week prior to first dose;
* Functional NENs which need to be treated with long acting Somatostatin analogues (SSAs) to control disease related syndromes, such as insulinoma, gastrinoma, glucagonoma, somatostatinoma, ACTHoma, VIPoma, accompanied by carcinoid syndrome, Zollinger-Ellison syndrome or other active symptoms;
* Previously treated with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CTLA-4 antibody, any other antibody acting on the T cell stimulation or checkpoint pathway or Surufatinib;
* Previously received anti-VEGF/VEGFR targeted drugs and progressed during the treatment or within 4 months after these drugs;
* Thyroid dysfunction with symptoms or require treatment when screening except hypothyroidism controlled only by thyroid hormone replacement therapy, the level of TSH in patients with iodine refractory differentiated thyroid cancer is more than 0.1 mU/L (or other corresponding unit level) before the beginning of the study treatment;
* Previously received immunosuppressive drugs except locally or temporarily used glucocorticoids;
* Autoimmune disease with systematic treatment or autoimmune disease history within 2 years;
* Previously received systematic immunologic stimulants within 4 weeks prior to the first dose;
* Inoculated with any live vaccine or attenuated live vaccine within 4 weeks or planed to inoculate during the study;
* Major surgery within 4 weeks or unhealed wound/fracture;
* Uncontrolled malignant hydrothorax, ascites, or pericardial effusion;
* Under anti-hypertension treatment, still uncontrolled hypertension, defined as: systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg;
* Disease or situation that affects drug absorption, or unable to take drugs orally;
* Previously received CYP3A4 strong inducers or strong inhibitors within 1 week or 5 half-life periods;
* Active gastric and duodenal ulcers, ulcerative colitis and other digestive disease, gastrointestinal tumor with active bleeding, or other gastrointestinal conditions that may cause bleeding or perforation by investigator's discretion;
* History or presence of a serious hemorrhage (>30 ml within 2 months), hemoptysis (>5 ml blood within 4 weeks) within 2 months;
* History or presence of an artery thrombosis or deep venous thrombosis within 6 months, or a thromboembolic event (including transient ischemic attack) within 12 months;
* Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction within 6 months prior to first dose, severe/unstable angina pectoris or coronary artery bypass grafting, congestive heart failure according to the New York Heart Association (NYHA) classification ≥ 2; ventricular arrhythmias which needs drug treatment; left ventricular ejection fraction (LVEF) <50%;
* Severe electrolyte abnormalities with clinical significance by investigator's discretion;
* Any clinically significant active infection, or unknown reason fever prior to first dose (temperature > 38.5℃);
* Active tuberculosis, on treatment or previously received antituberculosis therapy within 1 year;
* History or presence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia or severely injured lung function except radiation pneumonia in the radiotherapy area;
* A positive immunodeficiency virus (HIV) test;
* History of clinically significant hepatic disease, including, but not limited to, known hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×10^3/ml or > 200 IU/ml); known Hepatitis C virus (HCV) infection with HCV RNA positive (copies ≥1×10^3/ml); or liver cirrhosis, etc.;
* Previously received investigational treatments unlisted in China within 4 weeks prior to first dose;
* Women who are pregnant or lactating;
* Previously allergic to any of the JS001 or Surufatinib ingredients, or monoclonal antibody;
* Any other conditions are inappropriate for the use of the investigational products by investigator's discretion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) of safety run-in part | From Cycle 1 Day 1 to the end of Cycle 2 Day 7 (each cycle is 21 days)
  The AEs of the first 6 patients were evaluated by the possibly occurs Dose Limited Toxicity (DLT).
Objective response rate (ORR) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy(up to approximately 2 years)
  The incidence of confirmed complete response or partial response (RECIST1.1).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy(up to approximately 2 years)
  The incidence of confirmed complete response or partial response (irRECIST).
Duration of Response (DoR) (RECIST1.1 and irRECIST) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  Duration from the first time reported partial response or complete response to the first time of disease progression or death.
Progression-free Survival (PFS) (RECIST1.1 and irRECIST) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  A duration from the date of initial treatment with Surufatinib combined with Toripalimab to disease progression or death of any cause.
Disease Control Rate (DCR) (RECIST1.1 and irRECIST) | From date of first dose of study drug until disease progression, withdrawal of consent, death, new anti-cancer therapy (up to approximately 2 years)
  Proportion of patients whose tumor volume control (reduced or enlarged) reaches a predetermined value and can maintain a minimum time limit.
Overall Survival (OS) | From date of first dose of study drug until withdrawal of consent or death (up to approximately 2 years)
  Duration from the date of initial treatment with Surufatinib plus toripalimab to the date of death due to any cause.
The AEs of all population | For each participant, from the first participant first dose until 30 days after the last dose (up to approximately 2 years)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered an investigational product.Safety and tolerance evaluated by incidence, severity and outcomes of AEs
Anti-drug Antibody (ADA) of Toripalimab | half of hour predose of Toripalimab for Cycle 1, 2, 3, 4, 5 (each cycle is 21 days) and 30 days after the last dose
  Blood samples will be collected and analyzed. Serum ADA will be detected by using validated methods.
Plasma maximum Concentration (Cmax) | Surufatinib (Cycle 1 and 3): Day 1: predose;1, 2, 4, 8,12 and 24 hours postdose. Toripalimab (Cycle 1 and 3): predose; 0.5, 2, 6, 12,24,48,96,168,336 and 504 hours postdose
  Blood samples will be collected at the designated time points.Cmax is the highest concentration of drug in the blood that is measured after a dose.
The drug concentration-time curve (AUC) | Surufatinib (Cycle 1 and 3): Day 1: predose;1, 2, 4, 8,12 and 24 hours postdose. Toripalimab (Cycle 1 and 3): predose; 0.5, 2, 6, 12,24,48,96,168,336 and 504 hours postdose
  Plasma samples will be collected at the designated time points. AUC represents the overall amount of drug in the bloodstream after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang P, Chen Z, Shi S, Li Z, Ye F, Song L, Zhang Y, Yin F, Zhang X, Xu J, Cheng Y, Su W, Shi M, Fan S, Tan P, Zhong C, Lu M, Shen L. Efficacy and safety of surufatinib plus toripalimab, a chemotherapy-free regimen, in patients with advanced gastric/gastroesophageal junction adenocarcinoma, esophageal squamous cell carcinoma, or biliary tract cancer. Cancer Immunol Immunother. 2024 May 7;73(7):119. doi: 10.1007/s00262-024-03677-7. PMID 38713205
- [Derived] Zhang P, Shi S, Xu J, Chen Z, Song L, Zhang X, Cheng Y, Zhang Y, Ye F, Li Z, Yin F, Ji D, Gao H, Li Y, Chen W, Yang M, Weng D, Wu C, Ma Y, Sheng W, Zhao Y, Yin X, Shen W, Su W, Shi M, Fan S, Tan P, Xu Q, Lu M, Shen L. Surufatinib plus toripalimab in patients with advanced neuroendocrine tumours and neuroendocrine carcinomas: An open-label, single-arm, multi-cohort phase II trial. Eur J Cancer. 2024 Mar;199:113539. doi: 10.1016/j.ejca.2024.113539. Epub 2024 Jan 15. PMID 38237373